CLINICAL TRIAL: NCT01273623
Title: A Prospective, Single-Arm Study to Evaluate the Effects of the Jetstream G3 System on Calcified Peripheral Vascular Lesions
Brief Title: The Jetstream G3™ Calcium Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1139
Record Dates: First submitted 2010-12-20; First posted 2011-01-10 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-10

CONDITIONS: Peripheral Arterial Disease
Keywords: PAD, Peripheral Arterial Disease, Calcium, Atherectomy, Jetstream
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with PAD (Experimental): Patients with symptomatic peripheral vascular disease undergoing percutaneous intervention who have moderate to severe obstructive intraluminal calcium
  Interventions: Device: Jetstream Atherectomy System

INTERVENTIONS:
Device: Jetstream Atherectomy System — to perform atherectomy on calcified lesions

SUMMARY:
To investigate the treatment effects with the Jetstream G3 System in moderate to severely calcified peripheral artery disease in the common femoral, superficial femoral or popliteal arteries using intravascular ultrasound (IVUS).

ELIGIBILITY:
Inclusion Criteria:

1. The patient is ≥ 18 years of age.
2. Patient has claudication determined to be due to femoropopliteal lesion(s) requiring revascularization.
3. The target lesion(s) is/are located in the common femoral, superficial femoral or popliteal arteries.
4. The reference vessel lumen (proximal to target lesion) is ≥ 3.0mm.
5. The patient is an acceptable candidate for percutaneous intervention using the Jetstream G3 System in accordance with its labeled indications and instructions for use.
6. The patient has signed approved informed consent.
7. Moderate or severe vessel obstructive intraluminal calcification as demonstrated by IVUS and angiography.

Exclusion Criteria:

1. Patient has an uncontrollable allergy to nitinol, stainless steel or other stent materials or to contrast agent.
2. Patient is unable to take appropriate anti-platelet therapy.
3. Patient has no distal runoff vessels.
4. Deep wall calcium.
5. Interventional treatment is intended for in-stent restenosis at the peripheral vascular site.
6. Patient has target vessel with moderate or severe angulation (e.g., >30 degrees) or tortuosity at the treatment segment.
7. Patient has a history of coagulopathy or hypercoagulable bleeding disorder.
8. Patient is receiving hemodialysis or has impaired renal function (creatinine is > 2.5 mg/dl) at the time of treatment.
9. Patient has evidence of intracranial or gastrointestinal bleeding within the past 3 months.
10. Patient has had severe trauma, fracture, major surgery or biopsy of a parenchymal organ within the past 14 days.
11. Patient is pregnant or nursing a child.
12. Intended interventional treatment includes planned laser, brachytherapy or atherectomy procedure other than the Jetstream G3 System.

    -

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Davis, MD, Principal Investigator — St. John Hospital; Malcolm Foster, Principal Investigator — Mercy Medical Center; Venkatesh Ramaiah, MD, Principal Investigator — Arizona Heart Institute; Joseph Ricotta, MD, Principal Investigator — Emory University; Thomas Shimshak, MD, Principal Investigator — Wheaton Franciscan Healthcare
Locations (5):
- United States (5):
  - Arizona Heart Institute, Phoenix, Arizona
  - Emory University, Atlanta, Georgia
  - St. John Hopital, Detroit, Michigan
  - Mercy Medical Center, Knoxville, Tennessee
  - Wheaton Franciscan Healthcare, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Yin D, Maehara A, Shimshak TM, Ricotta JJ 2nd, Ramaiah V, Foster MT 3rd, Davis TP, Matsumura M, Mintz GS, Gray WA. Intravascular Ultrasound Validation of Contemporary Angiographic Scores Evaluating the Severity of Calcification in Peripheral Arteries. J Endovasc Ther. 2017 Aug;24(4):478-487. doi: 10.1177/1526602817708796. Epub 2017 May 15. PMID 28504047

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: subjects with calcified peripheral arterial lesions determined by intravascular ultrasound
Period: Overall Study
Arm/Group | Single Arm
Started | 55 (met angiographic criteria)
Completed | 26 (met IVUS criteria)
Not Completed | 29
Not completed — did not meet IVUS criteria | 29

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Luminal Area Change
Description: lumen area change as measured by intravascular ultrasound (IVUS)
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: mm^2
Groups:
- Pre-atherectomy: prior to Jetstream use
- Post-atherectomy: after Jetstream use and prior to adjunctive therapies
Arm/Group | Pre-atherectomy | Post-atherectomy
Number analyzed (Participants) | 26 | 26
mm^2 | 5.1 (2.8) | 8.3 (2.6)
Statistical Analysis 1: Comparison: Pre-atherectomy vs Post-atherectomy; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Adjunctive Therapy Use
Time Frame: Day 0
Measure: Number; unit: percentage of participants
Arm/Group | Study Participants
Number analyzed (Participants) | 26
percentage of participants
  Percutaneous Transluminal Angioplasty | 62
  Stent | 31
  Other devices or procedures | 8

3. Secondary Outcome: Residual Diameter Stenosis
Description: lumen diameter stenosis change post-atherectomy
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Study Participants
Number analyzed (Participants) | 26
percentage change | -37 (13)

ADVERSE EVENTS:
Time Frame: through 30 days
Arm/Group | Study Participants
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Participants (N=26)
Death (Surgical and medical procedures) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0)
Unplanned amputation (Surgical and medical procedures) | 0 (0)
Target lesion revascularization (Surgical and medical procedures) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less